CLINICAL TRIAL: NCT01062113
Title: A Randomized, Double-Blind, Multicenter, Comparative Study To Evaluate Efficacy And Safety Of An Additional Dose Of Celecoxib (YM177) In The Treatment Of Acute Pain After Oral Surgery Lateral Mandibular Impacted Third Molar Tooth Extraction
Brief Title: Study To Evaluate Efficacy And Safety Of An Additional Dose Of Celecoxib (YM177) In Patients With Post-Tooth Extraction Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3191200
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Results first posted 2012-11-19 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Pain
Keywords: Acute pain after oral surgery lateral mandibular Impacted third molar tooth extraction
MeSH Terms: conditions — Pain | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Celecoxib 400mg (Experimental)
  Interventions: Drug: Celecoxib
- Celecoxib 200mg (Experimental)
  Interventions: Drug: Celecoxib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celecoxib — Initial dose: Celecoxib 200mg tablet x 2 will be administrated during a period from 1 to 2 hours post lateral mandibular impacted third molar tooth extraction in subjects with "moderate pain" or "severe pain"rated as 45.0 mm or more on the VAS
  Arms: Celecoxib 400mg
Drug: Celecoxib — Additional dose: Celecoxib 200mg tablet x 1 will be administrated during a period from 5 to 12 hours post-initial dose of Celecoxib 400mg in subjects who require an additional analgesic dose for any pain
  Arms: Celecoxib 200mg
Drug: Placebo — Additional dose: Placebo (tablet) will be administrated during a period from 5 to 12 hours post-initial dose of Celecoxib 400mg in subjects who require an additional analgesic dose for any pain
  Arms: Placebo

SUMMARY:
To evaluate efficacy and safety of additional dose of celecoxib, as compared to placebo, in patients with post lateral mandibular impacted third molar tooth extraction pain.

ELIGIBILITY:
Inclusion Criteria:

Initial dose:

* 20 to 64 years
* Patients with undergoing mandibular impacted third molar tooth extraction accompanied by lateral bone removal and crown cutting
* Patients with pain that meets both of the following criteria
* Pain intensity (4-categorical): "moderate pain" or "severe pain"
* Pain intensity (VAS): 45.0 mm or more

Additional dose:

* Patients with pain that corresponds to "4. Agree" or "5. Strongly agree" as the answer to the "question about the pain intensity" during the period from 5 hours to 12 hours post-initial dose of the study drug

Exclusion Criteria:

* Patients with acute inflammatory findings in the oral cavity necessitating treatment
* Patients who are scheduled to receive general anesthesia and analgesics in the process of the eligible tooth extraction

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 255 (Actual)
Dates: Start 2010-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- Japan (22):
  - Jyuzen General Hospital, Niihama-shi, Ehime
  - Kyushu Dental College Hospital, Kitakyusyu-shi, Fukuoka
  - Bishinkai Medical Corporation Health Park Clinic, Takasaki-shi, Gunma
  - Kure Kyosai Hospital, Kure-shi, Hiroshima
  - Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Kagawa University Faculty of Medicine University Hospital, Kita-gun, Kagawa-ken
  - Tokai University Hospital, Isehara-shi, Kanagawa
  - Kumamoto Medical Center, Kumamoto, Kumamoto
  - Sendai Medical Center, Sendai, Miyagi
  - Maruko Central General Hospital, Ueda-shi, Nagano
  - Nagano National Hospital, Ueda-shi, Nagano
  - The Nippon Dental University Niigata Hospital, Niigata, Niigata
  - Osaka Dental University Hospital, Osaka, Osaka
  - Osaka Prefectural General Medical Center, Osaka, Osaka
  - Meikai University Hospital, Sakado-shi, Saitama
  - Shizuoka Medical Center, Sunto-gun, Shizuoka
  - Tochigi National Hospital, Utsunomiya, Tochigi
  - Tokai University Hachioji Hospital, Hachiouji-shi, Tokyo
  - Japan Red Cross Musashino Hospital, Musashino-shi, Tokyo
  - Showa University Dental Hospital, Ōta-ku, Tokyo
  - Kanto Medical Center NTT EC, Shinagawa-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo

REFERENCES:
- [Derived] Saito K, Kaneko A, Machii K, Ohta H, Ohkura M, Suzuki M. Efficacy and safety of additional 200-mg dose of celecoxib in adult patients with postoperative pain following extraction of impacted third mandibular molar: a multicenter, randomized, double-blind, placebo-controlled, phase II study in Japan. Clin Ther. 2012 Feb;34(2):314-28. doi: 10.1016/j.clinthera.2012.01.004. Epub 2012 Jan 28. PMID 22284900
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191200&StudyName=Study%20To%20Evaluate%20Efficacy%20And%20Safety%20Of%20An%20Additional%20Dose%20Of%20Celecoxib%20%28YM177%29%20In%20Patients%20With%20Post-Tooth%20Extraction%20Pain

RESULTS

PARTICIPANT FLOW:
Groups:
- Initial Dose Celecoxib 400 mg: Included the participants who received initial dose of celecoxib 400 mg only
- Additional Dose Celecoxib 200 mg: Included participants who received celecoxib 200 mg as an additional dose from 5 to 12 hours after the initial dose (celecoxib 400 mg).
- Additional Dose Placebo: Included participants who received placebo as an additional dose from 5 to 12 hours after the initial dose (celecoxib 400 mg).
Period: Overall Study
Arm/Group | Initial Dose Celecoxib 400 mg | Additional Dose Celecoxib 200 mg | Additional Dose Placebo
Started | 133 | 64 | 58
Completed | 93 | 42 | 27
Not Completed | 40 | 22 | 31
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lack of Efficacy | 38 | 22 | 31
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Initial Dose Celecoxib 400 mg | Additional Dose Celecoxib 200 mg | Additional Dose Placebo | Total
Number analyzed (Participants) | 133 | 64 | 58 | 255
Age, Customized [Number; unit: participants]
  < 18 years | 0 | 0 | 0 | 0
  Between 18 and 64 | 133 | 64 | 58 | 255
  >= 65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 39 | 36 | 139
  Male | 69 | 25 | 22 | 116

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Rate (Percentage) of Patient's Impression
Description: Patient's impression was assessed by self-report and was entered in the patient diary, based on the following categories: "Excellent", " Good", "Fair" and "Poor".
  Efficacy rate was calculated from the following formula, "The number of participants assessed as Excellent or Good" over "total participants" multiplied by 100.
Time Frame: 2 hours post-additional dose
Population: The full analysis set (FAS). This analysis set consisted of randomized participants who received the additional dose of the study drug and who were assessed for at least one efficacy endpoint after randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Additional Dose Celecoxib 200 mg | Additional Dose Placebo
Number analyzed (Participants) | 64 | 58
percentage of participants | 64.1 | 25.9
Statistical Analysis 1: Comparison: Additional Dose Celecoxib 200 mg vs Additional Dose Placebo; Test type: Superiority or Other; p < 0.0001, asymptotic z-test — The difference in the efficacy rates was tested using normal distribution at a significance level of 2-sided 5%. 2-sided 95% confidence interval (CI) for the difference in the efficacy rates was calculated using normal approximation; Risk Difference (RD) = 38.2, 95% CI 2-sided [20.3 to 56.1], Standard Error of Mean 9.1

2. Secondary Outcome: Number of Participants in Each Pain Intensity (PI) With 4 Categories
Description: Pain intensity was entered in the patient diary on the following categories: "No pain", "Mild pain", "Moderate pain" and "Severe pain".
Time Frame: 2 hours after additional dose
Population: The full analysis set (FAS), Baseline Observation Carried Forward (BOCF).
Measure: Number; unit: participants
Groups:
- Additional Dose Celecoxib 200mg: Included participants who received Celecoxib 200 mg as an additional dose from 5 to 12 hours after the initial dose (celecoxib 400 mg).
Arm/Group | Additional Dose Celecoxib 200mg | Additional Dose Placebo
Number analyzed (Participants) | 64 | 58
participants
  None | 11 | 3
  Mild | 34 | 24
  Moderate | 18 | 28
  Severe | 1 | 3

3. Secondary Outcome: Pain Intensity Measured by Visual Analog Scale (VAS)
Description: The Pain intensity was recorded on the 100 mm VAS in the patient diary, where 0 mm=no pain, 100 mm=unbearable maximal pain.
Time Frame: 2 hours post-additional dose
Population: The full analysis set (FAS), Baseline Observation Carried Forward (BOCF).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Additional Dose Celecoxib 200 mg | Additional Dose Placebo
Number analyzed (Participants) | 64 | 58
mm | 35.8 (25.5) | 51.9 (21.9)
Statistical Analysis 1: Comparison: Additional Dose Celecoxib 200 mg vs Additional Dose Placebo; Test type: Superiority or Other; p = 0.0003, t-test, 2 sided

4. Secondary Outcome: Differences in Pain Intensity (PI) Measured by VAS Among Participants
Description: The differences in PI were obtained by subtracting the PI at each time point from the Baseline PI score.
Time Frame: Pre-additional dose (baseline) and 2 hours post-additional dose
Population: The full analysis set (FAS), Baseline Observation Carried Forward (BOCF).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Additional Dose Celecoxib 200 mg | Additional Dose Placebo
Number analyzed (Participants) | 64 | 58
mm | 33.4 (24.2) | 12.3 (19.5)
Statistical Analysis 1: Comparison: Additional Dose Celecoxib 200 mg vs Additional Dose Placebo; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From informed consent to Day 28 postdose
Arm/Group | Initial Dose Celecoxib 400 mg | Additional Dose Celecoxib 200 mg | Additional Dose Placebo
Serious Adverse Events (participants affected / at risk) | 0/133 | 0/64 | 0/58
Other Adverse Events (participants affected / at risk) | 25/133 | 13/64 | 18/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Dose Celecoxib 400 mg (N=133) | Additional Dose Celecoxib 200 mg (N=64) | Additional Dose Placebo (N=58)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Beta 2 microglobulin increased (Investigations) | 7 | 5 | 9
Beta-N-acetyl-D-glucosaminidase increased (Investigations) | 4 | 1 | 5
Blood bilirubin increased (Investigations) | 4 | 3 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 1
Blood phosphorus decreased (Investigations) | 1 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 2
Blood urea increased (Investigations) | 0 | 0 | 1
Blood urine present (Investigations) | 1 | 0 | 0
Protein urine present (Investigations) | 0 | 1 | 1
Urobilin urine present (Investigations) | 1 | 1 | 1
White blood cell count increased (Investigations) | 1 | 1 | 2
Adenocarcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.